CLINICAL TRIAL: NCT02994303
Title: Podocyturia, a Non-Invasive Predictor of Renal Dysfunction in Fabry Nephropathy
Brief Title: Podocyturia - Predictor of Renal Dysfunction in Fabry Nephropathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Lysosomal Disease Network (Other)
Responsible Party: Principal Investigator, Behzad Najafian, Associate Professor, Director, Electron Microscopy Laboratory, University of Washington
Other Study IDs: 51316-EA; U54NS065768 (NIH)
Record Dates: First submitted 2016-12-05; First posted 2016-12-15 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Fabry Disease
Keywords: Fabry disease; Fabry nephropathy; end-stage renal disease; Anderson-Fabry disease; Fabry's disease
MeSH Terms: conditions — Fabry Disease; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine Sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In patients with Fabry disease, this research study explores the presence of podocytes in their urine as a potential non-invasive biomarker for baseline kidney disease; and explores changes in the quantity of podocytes in their urine over time as a predictor for kidney disease progression. To accomplish this, the investigators will evaluate the quantification of podocytes in the urine of Fabry disease patients at baseline and longitudinally over time. This study requires a single patient visit, during which the patient provides a urine specimen. The research team will then collect the patient's kidney function data proximate to the time of urine collection, and follow the patient's kidney function data longitudinally over the five years of this study by reviewing their medical charts. The study offers no interventions.

DETAILED DESCRIPTION:
Despite long-term recombinant enzyme replacement therapy, kidney failure remains a common and important complication of Fabry disease. Recent studies suggest that early administration of enzyme replacement therapy in sufficient dosage may prevent progression of kidney failure in patients with Fabry disease. Currently, there is no reliable non-invasive biomarker to detect early, occult kidney injury in these patients. Such early kidney injury detection is critical for guiding the decision as to when to initiate enzyme replacement therapy, and for identifying those patients with more severe kidney injury who may need higher doses of enzyme replacement therapy or additional forms of therapy.

Podocytes are special kidney cells with a crucial role in preventing escape of protein from the blood into the urine. Biopsy studies of Fabry disease patients suggest that podocyte injury occurs early and is progressive with increasing age in young Fabry disease patients. It is also likely that podocyte injury and loss leads to irreversible kidney lesions in later stages of Fabry disease nephropathy. Because injured podocytes are sloughed off into the urine (a manifestation known as podocyturia), quantification of urine podocytes might serve as a non-invasive and sensitive biomarker useful for predicting Fabry disease nephropathy risk; and to guide more effective Fabry disease treatment.

The investigators' preliminary data show correlations between presence of urinary podocytes and other markers of renal disease in adult Fabry disease patients; however, these cross-sectional data need to be expanded. The investigators have no information as to whether this potential biomarker could predict progression of the disease.

The investigators hypothesize that since podocyte injury plays a central role in kidney complications of Fabry disease, podocyte loss detected in the urine will identify patients with greater underlying kidney disease, and will identify patients with greater propensity for kidney disease progression. They also hypothesize that the number of podocytes in the urine of patients with Fabry disease will correlate directly with these patients' proteinuria, and will correlate inversely with their glomerular filtration rate (GFR) at baseline. Additionally the investigators hypothesize that the number of podocytes in the urine of patients with Fabry disease will predict increase in proteinuria and decline in glomerular filtration rate, as measured during long-term patient follow-up.

Data to be collected include identification of these patients' GLA gene mutation; measurement of their baseline a-galactosidase A enzyme activity; their baseline age, gender, height and weight; measurement of their baseline serum creatinine (SCr), eGFR, PCR and ACR; these patients' family history of Fabry disease, their history of kidney or systemic diseases, their medications including enzyme replacement therapy, and their medical information about other complications of Fabry disease (such as cardiomyopathy, arrhythmias, neuropathy and gastrointestinal problems).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been diagnosed with Fabry disease
* Patients must be between the ages of 1 day-90 years

Exclusion Criteria:

* Fabry disease patients who have had a renal transplant
* Fabry disease patients who are, or have been, subjects in any investigational drug study

Ages: 1 Day to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of any gender who have been diagnosed with Fabry disease
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2014-09; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Detection of Podocyturia in Subjects Diagnosed with Fabry Disease | At time of enrollment
  In subjects who have been diagnosed with Fabry disease, their urine sample will be examined for the presence of podocyturia at time of enrollment. If podocyturia is present, it will be quantified and recorded.

SECONDARY OUTCOMES:
Change from Baseline in Number of Urine Podocytes at Year 1, 2, 3, 4 and 5 | Annually at Year 1, Year 2, Year 3, Year 4 and Year 5
  For Fabry disease patients who tested positive at time of enrollment for the presence of urine podocytes, annually during the five years of this study their medical records will be used as the information source to record their numbers of urine podocytes. This annual podocyte-count data will be analyzed to determine whether change over time has occurred in their number of urine podocytes, and if it has occurred, to examine if this change correlates with changes in urine albumin excretion, urine protein excretion or glomerular filtration rate, as extracted from electronic medical records.
Change from Baseline in urine protein/creatinine ratio (PCR) at Year 1, 2, 3, 4 and 5 | At time of enrollment, then annually at Year 1, Year 2, Year 3, Year 4 and Year 5
  In patients who have been diagnosed with Fabry disease, their urine protein/creatinine ratio (PCR) will be quantified at time of enrollment; and annually thereafter for five years by collection of data from their medical chart. Their quantified podocyturia will be correlated with change in their urine protein/creatinine ratio (PCR) over time.
Change from Baseline in urine albumin/creatinine ratio (ACR) at Year 1, 2, 3, 4 and 5 | At time of enrollment, then annually at Year 1, Year 2, Year 3, Year 4 and Year 5
  In patients who have been diagnosed with Fabry disease, their urine albumin/creatinine ratio (ACR) will be quantified at time of enrollment; and annually thereafter for five years by collection of data from their medical chart. Their quantified podocyturia will be correlated with change in their urine albumin/creatinine ratio (ACR) over time.
Change from Baseline in estimated glomerular filtration rate (eGFR) at Year 1, 2, 3, 4 and 5 | At time of enrollment, then annually at Year 1, Year 2, Year 3, Year 4 and Year 5
  In patients who have been diagnosed with Fabry disease, their estimated glomerular filtration rate (eGFR) will be quantified at time of enrollment; and annually thereafter for five years by collection of data from their medical chart. Their quantified podocyturia will be correlated with change in their estimated glomerular filtration rate (eGFR) over time.
Change from Baseline in Number of Urine Podocytes at Year 1, 2, 3, 4 or 5, Based On Subject's New Urine Sample | Annually at Year 1, Year 2, Year 3, Year 4 or Year 5
  Providing more than one urine sample for podocyte counting is optional in this study. For those subjects who do provide an additional urine specimen in any year of this study that is subsequent to baseline, the number of urine podocytes at baseline will be compared to the number of urine podocytes in any additional urine specimen(s) collected in years 1 through 5. This podocyte-count data will be analyzed to determine whether change over time has occurred in their number of urine podocytes, and if it has occurred, to examine if this change correlates with changes in urine albumin excretion, urine protein excretion or glomerular filtration rate, as extracted from electronic medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Behzad Najafian, M.D., Principal Investigator — University of Washington Associate Professor, Pathology
Locations (3):
- United States (3):
  - Emory University, Decatur, Georgia
  - University of Minnesota, Minneapolis, Minnesota
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data is input to the NIH-funded Rare Diseases Clinical Research Network's Data Management & Coordinating Center ("DMCC"). Eventually this data will become part of the database of Genotypes and Phenotypes ("dbGaP"), which is part of the National Center for Biotechnology Information, U.S. National Library of Medicine.

REFERENCES:
- [Background] Najafian B, Tondel C, Svarstad E, Sokolovkiy A, Smith K, Mauer M. One Year of Enzyme Replacement Therapy Reduces Globotriaosylceramide Inclusions in Podocytes in Male Adult Patients with Fabry Disease. PLoS One. 2016 Apr 15;11(4):e0152812. doi: 10.1371/journal.pone.0152812. eCollection 2016. PMID 27081853
- [Background] Najafian B, Fogo AB, Lusco MA, Alpers CE. AJKD Atlas of Renal Pathology: Fabry nephropathy. Am J Kidney Dis. 2015 Nov;66(5):e35-6. doi: 10.1053/j.ajkd.2015.08.006. No abstract available. PMID 26498420
- [Background] Wijburg FA, Benichou B, Bichet DG, Clarke LA, Dostalova G, Fainboim A, Fellgiebel A, Forcelini C, An Haack K, Hopkin RJ, Mauer M, Najafian B, Scott CR, Shankar SP, Thurberg BL, Tondel C, Tylki-Szymanska A, Ramaswami U. Characterization of early disease status in treatment-naive male paediatric patients with Fabry disease enrolled in a randomized clinical trial. PLoS One. 2015 May 8;10(5):e0124987. doi: 10.1371/journal.pone.0124987. eCollection 2015. PMID 25955246
- [Background] Mauer M, Glynn E, Svarstad E, Tondel C, Gubler MC, West M, Sokolovskiy A, Whitley C, Najafian B. Mosaicism of podocyte involvement is related to podocyte injury in females with Fabry disease. PLoS One. 2014 Nov 11;9(11):e112188. doi: 10.1371/journal.pone.0112188. eCollection 2014. PMID 25386848
- [Background] Najafian B, Mauer M, Hopkin RJ, Svarstad E. Renal complications of Fabry disease in children. Pediatr Nephrol. 2013 May;28(5):679-87. doi: 10.1007/s00467-012-2222-9. Epub 2012 Aug 17. PMID 22898981
- [Background] Najafian B, Mauer M. Quantitating glomerular endothelial fenestration: an unbiased stereological approach. Am J Nephrol. 2011;33 Suppl 1(Suppl 1):34-9. doi: 10.1159/000327075. Epub 2011 Jun 10. PMID 21659733
- [Background] Najafian B, Svarstad E, Bostad L, Gubler MC, Tondel C, Whitley C, Mauer M. Progressive podocyte injury and globotriaosylceramide (GL-3) accumulation in young patients with Fabry disease. Kidney Int. 2011 Mar;79(6):663-670. doi: 10.1038/ki.2010.484. Epub 2010 Dec 15. PMID 21160462
- [Background] Ramaswami U, Najafian B, Schieppati A, Mauer M, Bichet DG. Assessment of renal pathology and dysfunction in children with Fabry disease. Clin J Am Soc Nephrol. 2010 Feb;5(2):365-70. doi: 10.2215/CJN.08091109. Epub 2010 Jan 7. PMID 20056758
- [Background] Mauer M, Najafian B. Implications of early renal changes in Fabry disease. Clin Ther. 2008;30 Suppl B:S40. doi: 10.1016/s0149-2918(08)80034-3. No abstract available. PMID 18395133
- [Background] Hopkin RJ, Cabrera G, Charrow J, Lemay R, Martins AM, Mauer M, Ortiz A, Patel MR, Sims K, Waldek S, Warnock DG, Wilcox WR. Risk factors for severe clinical events in male and female patients with Fabry disease treated with agalsidase beta enzyme replacement therapy: Data from the Fabry Registry. Mol Genet Metab. 2016 Sep;119(1-2):151-9. doi: 10.1016/j.ymgme.2016.06.007. Epub 2016 Jun 13. PMID 27510433
- [Background] Hopkin RJ, Jefferies JL, Laney DA, Lawson VH, Mauer M, Taylor MR, Wilcox WR; Fabry Pediatric Expert Panel. The management and treatment of children with Fabry disease: A United States-based perspective. Mol Genet Metab. 2016 Feb;117(2):104-13. doi: 10.1016/j.ymgme.2015.10.007. Epub 2015 Oct 23. PMID 26546059
- [Background] Warnock DG, Mauer M. Fabry disease: dose matters. J Am Soc Nephrol. 2014 Apr;25(4):653-5. doi: 10.1681/ASN.2013121322. Epub 2014 Feb 20. No abstract available. PMID 24556355
- [Result] Fall B, Scott CR, Mauer M, Shankland S, Pippin J, Jefferson JA, Wallace E, Warnock D, Najafian B. Urinary Podocyte Loss Is Increased in Patients with Fabry Disease and Correlates with Clinical Severity of Fabry Nephropathy. PLoS One. 2016 Dec 16;11(12):e0168346. doi: 10.1371/journal.pone.0168346. eCollection 2016. PMID 27992580
- See also: Web site of the University of Washington in Seattle, Washington. This is the location of this research study's Principal Investigator and his team. — http://www.washington.edu
- See also: Web site of Emory University, one of the satellite locations of this research study. — http://www.emory.edu/home/index.html
- See also: Web site of the University of Minnesota - Twin Cities, one of the satellite locations of this research study. — https://twin-cities.umn.edu/